CLINICAL TRIAL: NCT06402422
Title: Vulnerability Markers for Depression: a Concurrent TMS-fNIRS Study
Brief Title: Vulnerability Markers for Depression
Status: Completed | Type: Observational
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Dr Georg Kranz, Assistant Professor, The Hong Kong Polytechnic University
Other Study IDs: HSEARS20230705001
Record Dates: First submitted 2024-04-24; First posted 2024-05-07 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2024-12

CONDITIONS: Major Depressive Disorder Remission; Major Depressive Disorder; Healthy
Keywords: Theta-burst stimulation; Concurrent TBS/fNIRS; Verbal fluency task
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- rMDD patients: Participants are required to visit the lab twice. In the first visit, participants will first perform a verbal fluency task during which the brain activity will be recorded by fNIRS. Then participants complete a cognitive test called Raven's Advanced Progressive matrices (~ 40 min). In the second visit, participants will receive concurrent iTBS/fNIRS.
  Interventions: Device: Theta-burst stimulation
- MDD patients: Participants are required to visit the lab twice. In the first visit, participants will first perform a verbal fluency task during which the brain activity will be recorded by fNIRS. Then participants complete a cognitive test called Raven's Advanced Progressive matrices (~ 40 min). In the second visit, participants will receive concurrent iTBS/fNIRS.
  Interventions: Device: Theta-burst stimulation
- Health Controls: Participants are required to visit the lab twice. In the first visit, participants will first perform a verbal fluency task during which the brain activity will be recorded by fNIRS. Then participants complete a cognitive test called Raven's Advanced Progressive matrices (~ 40 min). In the second visit, participants will receive concurrent iTBS/fNIRS.
  Interventions: Device: Theta-burst stimulation
- High Risk-HCs: Participants are required to visit the lab twice. In the first visit, participants will first perform a verbal fluency task during which the brain activity will be recorded by fNIRS. Then participants complete a cognitive test called Raven's Advanced Progressive matrices (~ 40 min). In the second visit, participants will receive concurrent iTBS/fNIRS.
  Interventions: Device: Theta-burst stimulation

INTERVENTIONS:
Device: Theta-burst stimulation — TBS comprises 3-pulse 50-Hz bursts, applied every 200 ms (at 5 Hz). iTBS consists of 2-second trains with an inter-train interval of 8 seconds. The investigators will repeat the trains (30 pulses; 10 bursts) 20 times to reach a total number of 600 pulses (3x10x20). Concurrent iTBS/fNIRS stimulation will be applied over the left DLPFC at an intensity of 90% resting motor threshold (RMT). This corresponds to ~110% of the active motor threshold. Stimulation at 90% RMT will also ensure compliance, reduce sensory discomfort and minimize dropout rates. Still, scalp discomfort will be recorded directly after the stimulation. The stimulation site over the DLPFC will be determined using the international 10-20 system and correspond to the F3 label.
  Other Names: Repetitive transcranial magnetic stimulation (rTMS)

SUMMARY:
The current study is a pilot for the GRF project entitled "Predicting illness trajectories in fully remitted major depression using concurrent TBS/fNIRS". The project aims to determine whether immediate prefrontal excitability modulated by intermittent theta-burst stimulation (iTBS) is altered in remitted major depressive disorder (rMDD) and therefore classifies as a potential trait marker to predict the incidence of recurrence. In the present cross-sectional study, we will recruit four clusters of population, including patients diagnosed with rMDD, currently depressed patients with varying numbers of episodes, healthy subjects, and never-depressed healthy subjects with elevated risk for MDD (defined as having a first-degree relative with a history of depression), to investigate the relationship between the number of prior episodes, cognitive function, and TBS-induced instantaneous brain activity change in the presumed neuropathological prefrontal cortex (PFC).

ELIGIBILITY:
Inclusion Criteria:

* rMDD patients: (a) aged 18 to 65; (b) a clinical diagnosis of recurrent depressive disorder by an experienced psychiatrist but currently in full remission (ICD 11, 6A71.7) according to results of the Mini International Neuropsychiatric Interview (MINI) and the Patient Health Questionnaire (PHQ-9), with a score ≤ 4; (c) at least two previous MDEs within the last 10 years; (d) no or stable (≥4 weeks) psychopharmacological medication.

Current MDD patients: (a) aged 18 to 65; (b) a clinical diagnosis of current unipolar depressive disorder by an experienced psychiatrist according to DSM-IV; (c) no or stable (≥4 weeks) psychopharmacological medication.

HCs: (a) aged 18 to 65 and (b) healthiness based on history and psychiatric assessment.

never-depressed HCs with elevated risk for MDD (HR-HCs): (a) aged 18 to 65, (b) healthiness based on history and psychiatric assessment and (c) with a family history of psychiatric illnesses.

Exclusion Criteria:

* rMDD patients: (a) severe internal diseases; (b) neurological disorders or a history of severe head injuries; (c) current psychiatric comorbidities, including addiction; (d) pregnancy; (e) common fNIRS and TMS exclusion criteria, such as a history of brain surgery, head injury, cardiac pacemaker, deep brain stimulation, intracranial metallic particles, history of seizures, and antiepileptics and benzodiazepines corresponding to a dose of >1 mg lorazepam/d.

MDD patients: (a) severe internal diseases; (b) neurological disorders or a history of severe head injuries; (c) Axis-I disorders and history of alcohol or substance abuse or past co-morbid axis-I disorders being the likely primary cause of the depressive syndrome within the past 6 months; (d) pregnancy; (e) common fNIRS and TMS exclusion criteria, such as a history of brain surgery, head injury, cardiac pacemaker, deep brain stimulation, intracranial metallic particles, history of seizures, and antiepileptics and benzodiazepines corresponding to a dose of >1 mg lorazepam/d.

HCs: (a) medical history of a major systemic illness or a neurological or psychiatric disorder; (b) psychiatric disorders in their first-degree relatives; (c) pregnancy; and (d) common fNIRS and TMS exclusion criteria as stated above.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Four clusters of the population will be recruited, including patients diagnosed with rMDD, currently depressed patients with varying numbers of episodes, healthy subjects, and never-depressed healthy subjects with elevated risk for MDD (defined as having a first-degree relative with a history of depression)
Sampling Method: Non-Probability Sample
Enrollment: 166 (Actual)
Dates: Start 2023-10-08 (Actual); Primary Completion 2024-12-18 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Oxyhemoglobin (HbO) change compared to baseline | During and within 3 minutes post TBS-fNIRS measurement.
  Primary imaging outcome measure: iTBS-induced HbO change in the bilater prefrontal cortex during and after stimulation.
Verbal fluency task induced-oxyhemoglobin (HbO) change compared to baseline | During the 60 seconds word-generation blocks.
  Primary imaging outcome measure: cognitive task-induced HbO change in the bilateral prefrontal cortex.

CONTACTS AND LOCATIONS:
Overall Officials: Georg S Kranz, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
PD may be shared upon request
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Upon request
Access Criteria: Upon request